CLINICAL TRIAL: NCT02571738
Title: A Multicenter, Randomized, Single-Blind Study With an Open-Label Extension Option to Further Evaluate the Safety and Efficacy of Cryopreserved Human Amniotic Membrane for the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Study to Evaluate the Safety and Efficacy of CHAM* for the Treatment of Diabetic Foot Ulcers
Acronym: *OTI-15-01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company's desire to allocate more research and development resources to other clinical programs. Decision not driven by any safety concerns.
Sponsor: Osiris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Osiris Protocol 303
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Chronic Diabetic Foot Ulcers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHAM (Active Comparator): Cryopreserved Human Amniotic Membrane
  Interventions: Biological: CHAM
- Control (Placebo Comparator): Standard of Care
  Interventions: Other: Control

INTERVENTIONS:
Biological: CHAM — The treatment indication is for chronic diabetic foot ulcers that can accommodate up to one 5cm x 5cm piece of CHAM
  Arms: CHAM
Other: Control — Standard of Care
  Arms: Control

SUMMARY:
A Multicenter, Randomized, Single-Blind Study with an Open-Label Extension Option to Further Evaluate the Safety and Efficacy of Cryopreserved Human Amniotic Membrane for the Treatment of Chronic Diabetic Foot Ulcers

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 years and 80 years of age inclusive, as of the date of screening
2. Confirmed diagnosis of Type I or Type II Diabetes
3. An Index Ulcer defined as chronic (presence of wound for > 4 weeks), but not present for more than 52 weeks at the Screening Visit
4. Index Ulcer is located below the malleoli on the plantar or dorsal surface of the foot
5. The Index Ulcer is between 1 cm2 and 15 cm2, inclusive, at the Screening Visit
6. The Index Ulcer extends into the dermis or subcutaneous tissue without evidence of exposed muscle, tendon, bone, or joint capsule
7. Wound is free of necrotic debris
8. Patient has adequate circulation to the foot as documented by either:

   * Ankle Brachial Index (ABI) > 0.70 and < 1.30, or
   * In patients with non-compressible ankle vessels defined as an ABI ≥ 1.30, a Toe Brachial Index (TBI) ≥ 0.50, or
   * In patients with non-compressible ankle vessels defined as an ABI ≥ 1.30 and TBI cannot be performed (e.g., toe is absent, wounds are present, or site cannot perform a TBI), a Doppler waveform in the posterior tibial or dorsalis pedis arteries at the ankle consistent with adequate flow in the foot (biphasic or triphasic) and other diagnostic confirmation of adequate flow (e.g., duplex imaging, normal pulse volume recording [PVR] testing).

Exclusion Criteria:

1. Index Ulcer is of non-diabetic pathophysiology
2. Gangrene is present on any part of the affected foot
3. Index Ulcer is over an active Charcot deformity
4. The longest dimension of the Index Ulcer exceeds 5 cm at the Baseline Visit
5. Patient is currently receiving dialysis or planning to go on dialysis
6. Patient has had 2 or more previous disease-related amputations of the lower extremities
7. Patient has a glycated hemoglobin A1c (HbA1c) level of >10%
8. Chronic oral steroid use >7.5 mg daily for longer than 3 months at the time of screening
9. Patient is receiving IV corticosteroids, immunosuppressive or cytotoxic agents at the time of screening
10. Requiring intravenous (IV) antibiotics to treat the index wound infection at the time of screening
11. Patient has an ulcer within 5 cm of the Index Ulcer identified for study consideration
12. Patient is Human Immunodeficiency Virus (HIV) positive or has Acquired Immune Deficiency Syndrome (AIDS)
13. Current evidence of cellulitis, or other evidence of infection including fever or pus drainage from the wound site
14. Current evidence of osteomyelitis or history of osteomyelitis within 30 days of screening
15. Patient has active malignancy other than non-melanoma skin cancer
16. Patient's Index Ulcer has decreased by ≥20% during 1-week screening period
17. Patient's random blood sugar is >350 mg/dl at screening
18. Patient has untreated alcohol or substance abuse at the time of screening
19. Pregnant women and women who are breastfeeding
20. Patient is currently enrolled or participated in another investigational device, drug, or biological trial within 30 days of screening
21. Patient has had within the last 30 days, or is currently undergoing, or is planning for wound treatments with growth factors, living skin, dermal substitutes or other advanced biological therapies
22. Patient is an employee, or an immediate family member of an employee, of the sponsor company or site research staff conducting the study
23. Patients who have already been randomized in Protocol 303 at any center may not be considered for screening or for re-entry into the trial at any center, even after the end of their follow-up period
24. Patients with a history of poor compliance, or an unwillingness or inability to adhere to the requirements of the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Complete closure of the index wound, defined as 100% re-epithelialization as determined by the Investigator, by the End of Single-Blind Treatment Visit with follow-up confirmation of continued closure at 2 consecutive study visits 2 weeks apart | Up to 112 days after Baseline Visit

SECONDARY OUTCOMES:
Complete index wound closure by the End of Single-Blind Treatment Visit as defined by 100% re-epithelialization, as determined by the Investigator. | Up to 84 days after Baseline Visit
Time to initial wound closure among patients that receive CHAM versus those that receive control as measured by Kaplan-Meier analysis. | Up to 84 days after Baseline Visit
Proportion of patients receiving CHAM that achieve a 50% reduction or greater in wound size by Day 28 (± 3 days) versus those that receive control. | Up to 28 days after Baseline
Number of applications of CHAM versus control | Up to 77 days after Baseline
Percentage of patients who achieve complete wound closure, defined as 100% re-epithelialization as determined by the Investigator, who participate in the Open-Label Treatment Phase | Up to 91 days after Single-Blind Treatment Phase

OTHER OUTCOMES:
Wound re-occurrence for up to 3 months after initial wound closure in patients receiving CHAM versus control. | Up to 84 days after Single-Blind Treatment Phase
Number and types of Adverse Events (AE) and Serious Adverse Events (SAE) | Up to 84 days after Single-Blind Treatment Phase
Number of patients with worsening of wound defined by a 50% increase in wound size | Up to 84 days after Baseline
Change in Quality of Life from Baseline, as determined by the Cardiff Wound Impact Schedule (CWIS) | Up to 84 days after Baseline

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - SAVAHCS, Tucson, Arizona
  - ILD Research Center, Carlsbad, California
  - Center for Clinical Research, Castro Valley, California
  - Center for Clinical Research, San Francisco, California
  - Stanford University, Stanford, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Barry University Clinical Research, North Miami Beach, Florida
  - SSH, South Weymouth, Massachusetts
  - Ocean County Foot & Ankle Surgical Associates, Toms River, New Jersey
  - NSLIJHS, Lake Success, New York
  - UNC, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Orthopedics, Altoona, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - North Texas Podiatric Medicine and Surgery Associates, Dallas, Texas
  - Texas Gulf Coast Medical Group, Webster, Texas